CLINICAL TRIAL: NCT02986919
Title: A Phase 2 Study of CPI-0610, a Small Molecule Inhibitor of Bromodomain and Extra-Terminal (BET) Proteins, in Patients With Malignant Peripheral Nerve Sheath Tumors
Brief Title: Study of CPI-0610 in Patients With Malignant Peripheral Nerve Sheath Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 092016-074
Record Dates: First submitted 2016-11-21; First posted 2016-12-08 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Nerve Tumors
Keywords: Malignant peripheral Nerve Sheath Tumors (MPNST); Neurofibromatosis sarcoma
MeSH Terms: conditions — Peripheral Nervous System Neoplasms; Neurofibrosarcoma | interventions — CPI-0610

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPI-0610 Treatment (Experimental): CPI-0610 will be administered 200mg orally once a daily for 14 consecutive days followed by a 7-day break.
  Interventions: Drug: CPI-0610

INTERVENTIONS:
Drug: CPI-0610 — * Optional tumor biopsy will be obtained prior to Day 1 of CPI-0610 administration.
  * CPI-0610 will be administered 200mg orally once a daily for 14 consecutive days followed by a 7-day break. The 14 days of CPI-0610 dosing and the 7-day break together constitute 1 cycle of treatment. The dose will not be adjusted for body weight or body surface area.

SUMMARY:
Establish safety and toxicity profile and preliminary response rate of CPI-0610 in MPNST patients and correlate response with pharmacodynamics markers and BET inhibition.

DETAILED DESCRIPTION:
* Optional tumor biopsy will be obtained prior to Day 1 of CPI-0610 administration.
* CPI-0610 will be administered 200mg orally once a daily for 14 consecutive days followed by a 7-day break. The 14 days of CPI-0610 dosing and the 7-day break together constitute 1 cycle of treatment. The dose will not be adjusted for body weight or body surface area.
* Patients should be instructed to take their daily dose at approximately the same time of day. Each dose should be taken with a glass of water and consumed over as short a time as possible-e.g., within 5 minutes. Patients should be instructed to swallow the tablet whole and to not chew or cut them.
* Doses may be taken either with or without food.
* If vomiting occurs during the course of treatment, then no re-dosing of the patient is allowed before the next scheduled dose.
* If the patient forgets to take his/her daily morning dose, then he/she should take CPI-0610 within 6 hours after the missed dose. If more than 6 hours have passed, then that day's dose should be omitted, and the patient should resume treatment with the next scheduled dose.
* Repeat optional tumor biopsy will be obtained on day 8 of CPI-0610 treatment.

Toxicities and Dosing Delays/Dose Modifications During a cycle of treatment, CPI-0610 should continue to be administered as planned unless CTCAE grade 3-4 toxicities occur. In the case of CPI-0610-related neutropenia and/or thrombocytopenia, dosing as planned should continue as long as the ANC remains >0.5x109/L and the platelet count remains >25x109/L. Should either the ANC or platelet count fall below these values-become CTCAE grade 4-dosing with CPI-0610 should be interrupted. CPI-0610 dosing within the planned 14 days of treatment should not be resumed until the ANC is >0.75x109/L and the platelet count is >50x109/L. In addition, dosing within the cycle of treatment should not be resumed if the interruption has resulted in the omission of more than 2 of the planned 14 days of dosing. If it is possible to resume dosing within the planned 14 days of treatment, no attempt should be made to make up the missed doses of CPI-0610. If more than 2 of the planned 14 days of therapy have been omitted, then treatment should be resumed only with a new cycle of treatment, if the ANC>1x109/L and the platelet count >75x109/L. In addition, all other toxicities considered to be related to CPI-0610 must have resolved to CTCAE grade 1 or baseline. If the patient fails to meet the above-cited criteria for retreatment, then initiation of the next cycle of treatment should be delayed by one week. Following the additional week of no treatment, the next cycle may begin if the patient's ANC is>1x109/L and the platelet count is >75x109/L. In addition, all other toxicities considered to be related to CPI-0610 must have resolved to CTCAE grade 1 or baseline. If there are more than 28 days between the start of one cycle and the start of the next, the patient will no longer receive CPI-0610 therapy unless the patient's MPNST is stable or responding to therapy. Then consideration may be given to resuming treatment at a lower dose level to be discussed with Sponsor and Institutional Review Board (IRB). When a reduction in dose of CPI-0610 is required, no re-escalation of dose will be permitted.

Exceptions to the toxicity delay are CTCAE elevations in alkaline phosphatase and uric acid and <72 hours of grade 3 fatigue. When laboratory abnormalities form the basis of treatment decisions, they should be confirmed by repeated testing with a new blood sample or procedure. Optimal therapy for vomiting or diarrhea is based on physician preference with consideration of the prohibited medications listed in the appendix. G-CSF may be used to treat patients who have developed dose-limiting neutropenia, as per institutional guidelines, following discontinuation of CPI-0610 treatment. However, G-CSF may not be used during CPI-0610 administration or during the treatment break. Patients should not have dose reductions of CPI-0610 unless a grade 3-4 toxicity occurs and retreatment is not possible within the 28 day period. Then the patient is withdrawn from study unless the patient's MPNST has responded or stable on therapy. Then consideration may be given to resuming treatment at a lower dose level to be discussed with Sponsor and IRB. When a reduction in the dose of CPI-0610 is required, no re-escalation of dose will be permitted. Patients whose treatment is interrupted or permanently discontinued because of toxicities must be followed until the toxicity resolves or stabilizes.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Must have histologically confirmed diagnosis of MPNST
3. Must have measurable disease by CT scan or MRI
4. Eastern Cooperative Oncology Group - ECOG performance status <2
5. Adequate organ and marrow function as defined below:

   * absolute neutrophil count greater than or equal to 1,000/mcL
   * platelets greater than or equal to 75,000/mcL
   * total bilirubin <2X normal institutional limits
   * AST(SGOT)/ALT(SPGT) greater than or equal to 2.5 X institutional upper limit of normal
   * creatinine <2X institutional upper limit of normal
6. Patients must have fully recovered from major surgery and from the acute toxic effects of prior chemotherapy and radiotherapy - residual grade 1 toxicity, e.g., grade 1 peripheral neuropathy and residual alopecia are allowed.
7. Female patients who are pre-menopausal or have experienced menopause for less than 2 years must have a negative serum pregnancy test <72 hours before starting study treatment. Male and female patients with reproductive potential must agree to use appropriate contraceptive methods while on study and for 3 months after the last dose of CPI-0610. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. Current infection with HIV, hepatitis B or hepatitis C. Patients will have serologic testing performed during screening for HIV and hepatitis B and C. Any serologic results suggestive of an ongoing viral infection will be further investigated as necessary to clarify the patient's status.
2. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of CPI-0610, including any unresolved nausea, vomiting, or diarrhea that is CTCAE grade >1.
3. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   Acute myocardial infarction or angina pectoris <6 months prior to starting study drug
4. Uncontrolled cardiac arrhythmia - patients with rate-controlled atrial fibrillation are not excluded.
5. A past medical history of other clinically significant cardiovascular disease - e.g., uncontrolled hypertension, history of labile hypertension or history of poor compliance with an antihypertensive regimen.
6. Any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study - e.g., clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection.
7. Systemic anti-cancer treatment or radiotherapy less than 2 weeks before the first dose of CPI-0610.
8. Treatment with an investigational small molecule less than 2 weeks before the first dose of CPI-0610.
9. Immunosuppressive treatment that cannot be discontinued prior to study entry and for the duration of the study. Immunosuppressive treatment should be discontinued for at least 1 week prior to start of the administration of CPI-0610. Oral prednisone at a dose of 10mg or less per day is allowed, as are other oral corticosteroids given at glucocorticoid-equivalent doses. Topical, nasal and inhaled corticosteroids are also allowed.
10. Pregnant or lactating women.
11. Women of child bearing potential and men with reproductive potential, if they are unwilling to use adequate contraception while on study therapy and for 3 months thereafter.
12. Use of strong CYP inhibitors or drugs that carry a definite risk of Torsades de Pointes.
13. Patients unwilling or unable to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Response rate of CPI-0610 | 21 day cycles for 84 days
  Establish the response rate of CPI-0610 in MPNST patients
Duration of CPI-0610 | 21 day cycles for 84 days
  Establish the response duration of CPI-0610 in MPNST patients
Adverse events associated with CPI-0610 | 21 day cycles for 84 days
  Describe the adverse events associated with CPI-0610 at the RP2D

SECONDARY OUTCOMES:
Correlate tumor exposure to CPI-0610 with tumor BIM1 expression | 21 day cycles for 84 days
  Correlate tumor exposure to CPI-0610 with tumor BIM1 expression

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No